CLINICAL TRIAL: NCT01271062
Title: Restoration of Beta Cell Function and Cardiovascular Parameters in Relation to Adipoinsular and Enteroinsular Axes After Gastric Bypass Surgery in Severely Obese Patients With Type 2 Diabetes
Brief Title: Restoration of Beta Cell Function and Cardiovascular Parameters in Relation to Adipoinsular and Enteroinsular Axes After Gastric Bypass Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cantonal Hospital of St. Gallen (Other)
Collaborators: European Foundation for the Study of Diabetes (Other); Medical University of Graz (Other)
Responsible Party: Principal Investigator, Bernd Schultes, Head of Interdisciplinary Obesity Center, Cantonal Hospital of St. Gallen
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: EKSG 09/061/2B
Record Dates: First submitted 2011-01-05; First posted 2011-01-06 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Diabetes Mellitus, Type 2; Bariatric Surgery Candidate
Keywords: Resolvment of Diabetes Mellitus, Type 2; gastric bypass
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- T2DM patients before gastric bypass surgery (Active Comparator): oral glucose tolerance test , botnia clamp, preoperative as well as 10 days postoperative and 1 year postoperative, gastric bypass surgery.
  Interventions: Procedure: gastric bypass surgery
- Non-diabetic patient before gastric bypass surgery (Active Comparator): oral glucose tolerance test , botnia clamp, preoperative as well as 10 days postoperative and 1 year postoperative, gastric bypass surgery.
  Interventions: Procedure: gastric bypass surgery
- non diabetic patients, non-bariatric abdominal surgery (Active Comparator): oral glucose tolerance test , botnia clamp, elective laparoscopic abdominal surgery.
  Interventions: Procedure: abdominal surgery
- severely obese T2DM patients following a very low caloric diet (Active Comparator): oral glucose tolerance test , botnia clamp, before as well after following a very low caloric diet. Very low caloric diet.
  Interventions: Behavioral: very low caloric diet

INTERVENTIONS:
Procedure: gastric bypass surgery
  Arms: Non-diabetic patient before gastric bypass surgery; T2DM patients before gastric bypass surgery
Procedure: abdominal surgery
  Arms: non diabetic patients, non-bariatric abdominal surgery
Behavioral: very low caloric diet
  Arms: severely obese T2DM patients following a very low caloric diet

SUMMARY:
Bariatric operations such as the gastric bypass procedure provide a unique in vivo model of improvement of pathological beta cell function. The presented double-centre study aims to comprehensively investigate different aspects of beta cell function in patients with type 2 diabetes (T2DM) with a wide range of disease duration after gastric bypass. In parallel, our project will address the aspects of changes in enteroinsular and adipoinsular axes as well as the early and late changes of other defined parameters after gastric bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* indication forbariatric surgery or non-bariatric abdominal surgery

Exclusion Criteria:

* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2009-10; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Acute insulin response (AIR) to glucose during IVGTT will be used as a primary variable characterizing the beta cell function | 10 days after gastric bypass

SECONDARY OUTCOMES:
OGTT calculations and modelling describing beta cell response to oral glucose load; Insulin and C-peptide areas under the curve (AUCs) during OGTT quantifying the incretin effect. | 10 days after gastric bypass
• Plasma concentrations and adipose tissue expression of selected adipokines and inflammatory cytokines characterizing the adipoinsular axis | 10 days after gastric bypass

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Schultes, Prof., Principal Investigator — Interdisciplinary Obesity Center, Kantonal Hospital St. Gallen, Switerland; Thomas Pieber, Prof., Principal Investigator — Division of Endocrinology and Nuclear Medicine, Department of Internal Medicine, Medical University of Graz, Austria
Locations (2):
- Division of Endocrinology and Nuclear Medicine, Department of Internal Medicine, MEdical University of Graz, Austria, Graz, Austria
- Interdisciplinary Obesity Center, Kantonal Hospital St. Gallen, Switzerland, Sankt Gallen, Switzerland